CLINICAL TRIAL: NCT03525158
Title: Intrusive Memories of Trauma Experienced by Young Refugees: Using Single Case Experimental Design to Investigate a Brief Cognitive Intervention Involving Computer Gameplay
Brief Title: A Brief Cognitive Intervention After Intrusive Memories of Trauma With Young Refugees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emily Holmes, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017/978-31
Record Dates: First submitted 2018-04-12; First posted 2018-05-15 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Intrusive Memories of Trauma, Symptom of Post Traumatic Stress Disorder (Criterion B1)

STUDY DESIGN:
Intervention Model Description: Single case experimental AB design with or without optional replication (ABAB) (ie no random assignment)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseline phase ('A') and Intervention phase ('B') (Other): Baseline phase ('A'): Measurements collected in a pen-and-paper diary four times a day (morning, afternoon, evening and night) over one week for the primary outcome (occurrence of intrusive memories of trauma). Individual baseline phases will be used as control periods.
  Intervention phase ('B'): A one-session intervention with a researcher including a simple cognitive task (a memory cue, 10 minutes time gap and ca. 20 minutes of Tetris game-play) followed by instructions to engage in the task self-guided over the subsequent week. Measurements collected in a pen-and-paper diary four times a day over one week following the intervention for the primary outcome (occurrence of intrusive memories of trauma).
  Interventions: Behavioral: Brief cognitive intervention

INTERVENTIONS:
Behavioral: Brief cognitive intervention — A one-session intervention with a researcher including a simple cognitive task (a memory cue, 10 minutes time gap and ca. 20 minutes of Tetris game play) with instructions to engage in the task self-guided in the subsequent week.

SUMMARY:
This research study is designed to investigate the use of a simple cognitive task (a memory cue and 10 minute time gap, followed by playing the computer game "Tetris") for decreasing the number of intrusive memories of trauma among young refugees and asylum seekers. The design is a single case experimental AB design with or without optional replication (ABAB). Participants will aim to complete a no-intervention phase ('A': baseline phase) of one week followed by a one-week intervention phase ('B'), including a one-session intervention with a researcher comprising the simple cognitive task, followed by instructions to continue to use the technique self-guided in the subsequent week. Follow ups are conducted after each week to monitor the occurrence of intrusive memories of trauma in a pen-and-paper diary. It is predicted that participants will report fewer intrusive memories during the intervention phase than during the preceding baseline phase.

ELIGIBILITY:
Inclusion Criteria:

* Refugee or asylum seeker
* Experiencing intrusive memories of trauma
* Have access to a smartphone
* Able to speak or read the study material in Swedish, English or Arabic
* Able to attend three meetings with a researcher

Exclusion Criteria:

* Exhibit psychotic symptoms or other symptoms of severe mental illness

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Change in the occurrence of intrusive memories of trauma from baseline week to intervention week | Baseline week 1 and Intervention week 1
  Number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) for one week during the baseline phase and one week during the intervention phase.

SECONDARY OUTCOMES:
Feasibility and acceptability ratings for using a smartphone game-play intervention | Intervention week 1
  Feasibility and Acceptability of the intervention was assessed with 10 self-rated items, e.g. "Would you recommend playing Tetris to a friend?". Scores could range from 0 - 10 with higher scores indicating greater acceptability/feasibility. Two items had open-ended follow-up questions: "How did you feel about playing Tetris after you had an intrusive memory?" and "Why"? or "How much would you prefer an intervention that is delivered by a computer/smartphone compared to seeing a doctor/psychologist in person?" and "Why"?
Self-guided intervention adherence - usage of the gameplay intervention in daily life | Intervention week 1
  Usage of the gameplay intervention was assessed with 4 self-rated items: 1. Did you play Tetris in the last week since the last meeting? (Yes/No). 2. If yes, how many days did you play Tetris in the last week since we first practiced the game together? 3. How long did you spend playing Tetris at a time? (<10 min - >30 min), 4. How often did you manage to play Tetris after you experienced an intrusive memory? (11-point scale; 0 = not at all; 10 = every time).
Impact of intrusive memories on concentration, control, sleep and stress | Baseline week 1 and Intervention week 1
  7 self-rated items were used to assess the impact of intrusive memories on concentration, control, sleep and stress: 2 items assessed experienced concentration difficulties due to intrusive memories and in general (11-point scale; high scores indicating more concentration difficulties); 1 item assessed for how long intrusive memories disrupted concentration (<1 min - >60 min), 1 item assessed feeling of control over intrusive memories (11-point scale, 0 = no control; 10 = in full control); 2 items assessed sleep disturbances due to intrusive memories (11-point scale; higher scores indicating more sleep disturbance); and 1 item assessed to what degree intrusive memories affected stress levels (11-point scale, 0 = not at all; 10 = affected very much). Two open-ended questions were included: "How do intrusive memories interfere with your concentration?" and "How do intrusive memories interfere with your ability to settle in to this country and learn new skills, such as a new language?"

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Prof, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Residental care home for young people, Stockholm
  - Swedish Language Classes for Refugees, Stockholm